CLINICAL TRIAL: NCT03097263
Title: Is the Walking Velocity an Efficient Outcome of Rehabilitation Program in Non- Specific Low Back Pain Patient
Acronym: MARLO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: CASILLAS Marlo 2016
Record Dates: First submitted 2016-11-03; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Non-specific Low Back Pain; Functional Capacities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients: Patients included for rehabilitation program
  Interventions: Other: Physical Rehabilitation program

INTERVENTIONS:
Other: Physical Rehabilitation program

SUMMARY:
Despite the prevalence of chronic low back pain, functional symptomatology of this disease remains poor and treatment decisions are based mainly on subjective data (importance and pain tolerance). However, there are some experimental elements that involve objective assessment of locomotor capabilities - at forefront objectives which the walking velocity in the evaluation of this pathology in terms of severity of functional impairment. Recent evidence suggest the effectiveness of physical rehabilitation program for improving patients functional capacities and their reintegration in socio-professional life. This retrospective study aims to quantify the evolution of the parameters collected during standardized walking tests performed before and after rehabilitation program. These patients have systematically carry out a comfortable walk test (400m walk test) and a brisk walk test (200m) at the beginning and end of their program. Furthermore, a maximal stress test on a treadmill was performed before the program in order to detect any cardiovascular events and to allow the personalization of the effort level required (target heart rate) during rehabilitation. In this study the evolution of the comfortable and fast speed will be collected and compared with the stress test data, and other measured parameters (functional score of Quebec, muscle Tests Shirado and Sorensen).

ELIGIBILITY:
Inclusion Criteria:

* Female or male
* age between 18 and 70
* Non-specific low back pain - achieved rehabilitation program

Exclusion Criteria:

* inflammatory diseases
* cancer
* infectious diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-specific low back pain patients included for rehabilitation program
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
COMFORTABLE WALKING SPEED (TEST OF 400M) | 4 weeks

SECONDARY OUTCOMES:
200m fast walk test walking velocity | 4 weeks
Quebec score | 4 weeks
Shirado test | 4 weeks
Sorensen test | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabiltiation department CHU Dijon, Dijon, France